CLINICAL TRIAL: NCT03231202
Title: A Multi-centre, Prospective, Randomized Controlled Study to Compare Outcomes of Non-operative Management (NOM) With and Without Splenic Arterial Embolization (SAE) in Hemodynamically Stable OIS Grade 4 and 5 Splenic Injuries.
Brief Title: Splenic Injury Embolization - the Question About NOM (SInE Qua NOM)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Christine Gaarder, Head, Department of Traumatology, Oslo University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2016/15608
Record Dates: First submitted 2017-07-05; First posted 2017-07-27 (Actual); Last update posted 2017-07-27 (Actual); Status verified 2017-07

CONDITIONS: Wounds and Injuries
Keywords: Non-operative management; Splenic Injury; Blunt; Splenic artery embolization; Trauma
MeSH Terms: conditions — Wounds and Injuries | interventions — Embolization, Therapeutic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Embolization (Experimental): The intervention arm will perform SAE as a central embolization of the splenic artery.
  Additional peripheral embolization is left to the discretion of the interventional radiologist.
  The study does not interfere with local diagnostic work-up and treatment protocols.
  Interventions: Procedure: Embolization
- Observation (No Intervention): The control arm in this randomized controlled trial will include only NOM patients diagnosed with splenic injuries OIS grade 4 or 5 and suitable for observation alone, and will comprise clinical observation according to local routines and protocols.

INTERVENTIONS:
Procedure: Embolization — The intervention arm will perform SAE as a central embolization of the splenic artery.
  Additional peripheral embolization is left to the discretion of the interventional radiologist.
  Other Names: Splenic artery embolization (SAE)
  Arms: Embolization

SUMMARY:
The primary objective is to compare the failure rate due to splenic bleeding between the patients undergoing pre-emptive splenic arterial embolization (SAE) as part of non-operative management (NOM) and the patients not undergoing SAE. We hypothesize that the use of pre-emptive SAE will decrease the delayed bleeding rate and increase the success rate of NOM.

DETAILED DESCRIPTION:
This randomised controlled study will follow the clinical course of hemodynamically normal trauma patients with Organ Injury Scale (OIS) grade 4 or 5 blunt splenic injuries, undergoing SAE or observation only until day 7 post injury. Only hemodynamically normal patients will be considered for enrolment into the study, and written informed consent from the patient is required.

CONTROL The control arm in this randomized controlled trial will include only NOM patients diagnosed with splenic injuries OIS grade 4 or 5 and suitable for observation alone, and will comprise clinical observation according to local routines and protocols. The patients will be observed with special focus on delayed bleeding and failure of NOM. A contrast enhanced US or CT scan with arterial phase will be performed on day 3-5 to exclude PSA. On day 7, the decision to perform SAE, splenectomy or continue NOM is left to the discretion of each participating institution, and registered in the case report form (CRF).

INTERVENTION The intervention arm will perform SAE as a central embolization of the splenic artery.

Additional peripheral embolization is left to the discretion of the interventional radiologist.

Each institution decides whether patients in the SAE group are to undergo immunization or not. The study does not interfere with local diagnostic work-up and treatment protocols.

We hypothesize that the use of pre-emptive SAE will decrease the delayed bleeding rate and increase the success rate of NOM leading to fewer splenectomies in this group of patients without concomitant increased complication rates. Additionally, we want to explore the effects of pre-emptive SAE vs observation alone on all cause failure rate, operative procedures, repeat angiography rate, complications, critical care stay, and mortality.

ELIGIBILITY:
Inclusion Criteria:

* blunt splenic injury OIS grade 4 or 5
* Adult trauma patients (according to local definitions)
* Present hemodynamically normal as judged by the responsible trauma consultant surgeon and eligible for NOM
* Randomised within 48 hours of injury
* Written informed consent is obtained

Exclusion Criteria:

* Hemodynamically compromised (not suitable for NOM)
* Needing transfusions
* CT shows evidence of significant contrast extravasation
* Other indications for laparotomy
* Prisoners
* Pregnant
* >80 years old
* Penetrating injury
* Contraindication to iv contrast

Ages: 16 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 224 (Estimated)
Dates: Start 2017-07-01 (Actual); Primary Completion 2019-08-01 (Estimated); Study Completion 2019-08-01 (Estimated)

PRIMARY OUTCOMES:
Failure of NOM | 7 days
  The primary objective is to compare the failure rate due to splenic bleeding between the patients undergoing pre-emptive SAE as part of NOM and the patients not undergoing SAE. The primary endpoint is the proportion of subjects failing NOM due to spleen related bleeding within 7 days of injury. All analyses will be based on an intention to treat analysis.

SECONDARY OUTCOMES:
Delayed bleeding episode | 6-12 weeks
  Incidence. Delayed bleeding episode is defined as hemodynamically unstable patient, CT verified contrast blush or drop in hemoglobin/hematocrit.
All cause and spleen related mortality | 6-12 weeks
  Incidence
All cause and spleen related failure of NOM | 6-12 weeks
  Incidence
Pseudoaneurysms (PSA) | 6-12 weeks
  Incidence
Symptomatic thromboembolic events | 6-12 weeks
  Incidence
Other spleen related complications | 6-12 weeks
  Incidence
Angiography related complications | 6-12 weeks
  Incidence

CONTACTS AND LOCATIONS:
Overall Officials: Christine Gaarder, MD, PhD, Principal Investigator — Head, Department of Traumatology
Locations (12):
- United States (3):
  - Denver Health Medical Center, Denver, Colorado
  - University of Pittsburgh School of Medicine, Pittsburgh, Pennsylvania
  - Harborview Medical Center, Seattle, Washington
- Liverpool Hospital, Sydney, Australia
- McGill University Health Centre, Montreal, Canada
- Rigshospitalet, Copenhagen, Denmark
- Kliniken der Stadt Köln, Cologne, Germany
- University Medical Center, Utrecht, Netherlands
- Oslo Universtity Hospital, Oslo, Norway
- Karolinska Institute, Stockholm, Sweden
- United Kingdom (2):
  - Royal London Hospital, London
  - Nottingham University Hospital, Nottingham

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Stassen NA, Bhullar I, Cheng JD, Crandall ML, Friese RS, Guillamondegui OD, Jawa RS, Maung AA, Rohs TJ Jr, Sangosanya A, Schuster KM, Seamon MJ, Tchorz KM, Zarzuar BL, Kerwin AJ; Eastern Association for the Surgery of Trauma. Selective nonoperative management of blunt splenic injury: an Eastern Association for the Surgery of Trauma practice management guideline. J Trauma Acute Care Surg. 2012 Nov;73(5 Suppl 4):S294-300. doi: 10.1097/TA.0b013e3182702afc. PMID 23114484
- [Result] Velmahos GC, Zacharias N, Emhoff TA, Feeney JM, Hurst JM, Crookes BA, Harrington DT, Gregg SC, Brotman S, Burke PA, Davis KA, Gupta R, Winchell RJ, Desjardins S, Alouidor R, Gross RI, Rosenblatt MS, Schulz JT, Chang Y. Management of the most severely injured spleen: a multicenter study of the Research Consortium of New England Centers for Trauma (ReCONECT). Arch Surg. 2010 May;145(5):456-60. doi: 10.1001/archsurg.2010.58. PMID 20479344
- [Result] Davis KA, Fabian TC, Croce MA, Gavant ML, Flick PA, Minard G, Kudsk KA, Pritchard FE. Improved success in nonoperative management of blunt splenic injuries: embolization of splenic artery pseudoaneurysms. J Trauma. 1998 Jun;44(6):1008-13; discussion 1013-5. doi: 10.1097/00005373-199806000-00013. PMID 9637156
- [Result] Schurr MJ, Fabian TC, Gavant M, Croce MA, Kudsk KA, Minard G, Woodman G, Pritchard FE. Management of blunt splenic trauma: computed tomographic contrast blush predicts failure of nonoperative management. J Trauma. 1995 Sep;39(3):507-12; discussion 512-3. doi: 10.1097/00005373-199509000-00018. PMID 7473916
- [Result] McIntyre LK, Schiff M, Jurkovich GJ. Failure of nonoperative management of splenic injuries: causes and consequences. Arch Surg. 2005 Jun;140(6):563-8; discussion 568-9. doi: 10.1001/archsurg.140.6.563. PMID 15967903
- [Result] Sclafani SJ, Weisberg A, Scalea TM, Phillips TF, Duncan AO. Blunt splenic injuries: nonsurgical treatment with CT, arteriography, and transcatheter arterial embolization of the splenic artery. Radiology. 1991 Oct;181(1):189-96. doi: 10.1148/radiology.181.1.1887032.
- [Result] Miller PR, Chang MC, Hoth JJ, Mowery NT, Hildreth AN, Martin RS, Holmes JH, Meredith JW, Requarth JA. Prospective trial of angiography and embolization for all grade III to V blunt splenic injuries: nonoperative management success rate is significantly improved. J Am Coll Surg. 2014 Apr;218(4):644-8. doi: 10.1016/j.jamcollsurg.2014.01.040. Epub 2014 Jan 28. PMID 24655852
- [Result] Bhullar IS, Frykberg ER, Siragusa D, Chesire D, Paul J, Tepas JJ 3rd, Kerwin AJ. Selective angiographic embolization of blunt splenic traumatic injuries in adults decreases failure rate of nonoperative management. J Trauma Acute Care Surg. 2012 May;72(5):1127-34. doi: 10.1097/TA.0b013e3182569849. PMID 22673236
- [Result] Schimmer JA, van der Steeg AF, Zuidema WP. Splenic function after angioembolization for splenic trauma in children and adults: A systematic review. Injury. 2016 Mar;47(3):525-30. doi: 10.1016/j.injury.2015.10.047. Epub 2015 Nov 19. PMID 26772452
- [Result] Haan JM, Bochicchio GV, Kramer N, Scalea TM. Nonoperative management of blunt splenic injury: a 5-year experience. J Trauma. 2005 Mar;58(3):492-8. doi: 10.1097/01.ta.0000154575.49388.74. PMID 15761342
- [Result] Skattum J, Titze TL, Dormagen JB, Aaberge IS, Bechensteen AG, Gaarder PI, Gaarder C, Heier HE, Naess PA. Preserved splenic function after angioembolisation of high grade injury. Injury. 2012 Jan;43(1):62-6. doi: 10.1016/j.injury.2010.06.028. Epub 2010 Jul 31. PMID 20673894
- [Result] Peitzman AB, Harbrecht BG, Rivera L, Heil B; Eastern Association for the Surgery of Trauma Multiinstitutional Trials Workgroup. Failure of observation of blunt splenic injury in adults: variability in practice and adverse consequences. J Am Coll Surg. 2005 Aug;201(2):179-87. doi: 10.1016/j.jamcollsurg.2005.03.037. PMID 16038813
- [Result] Cirocchi R, Boselli C, Corsi A, Farinella E, Listorti C, Trastulli S, Renzi C, Desiderio J, Santoro A, Cagini L, Parisi A, Redler A, Noya G, Fingerhut A. Is non-operative management safe and effective for all splenic blunt trauma? A systematic review. Crit Care. 2013 Sep 3;17(5):R185. doi: 10.1186/cc12868. PMID 24004931
- [Result] Zarzaur BL, Vashi S, Magnotti LJ, Croce MA, Fabian TC. The real risk of splenectomy after discharge home following nonoperative management of blunt splenic injury. J Trauma. 2009 Jun;66(6):1531-6; discussion 1536-8. doi: 10.1097/TA.0b013e3181a4ed11. PMID 19509611
- [Result] Clancy AA, Tiruta C, Ashman D, Ball CG, Kirkpatrick AW. The song remains the same although the instruments are changing: complications following selective non-operative management of blunt spleen trauma: a retrospective review of patients at a level I trauma centre from 1996 to 2007. J Trauma Manag Outcomes. 2012 Mar 13;6(1):4. doi: 10.1186/1752-2897-6-4. PMID 22410104